CLINICAL TRIAL: NCT03387709
Title: Effects of Pistachio Consumption in a Weight Loss Intervention on Weight Change, Dietary Intake and Metabolic Factors
Brief Title: UCSD Get Fit, Be Fit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American Pistachio Growers (Other)
Responsible Party: Principal Investigator, Cheryl Rock, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 172109
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Overweight and Obesity
Keywords: Nondiabetic; Overweight; Obesity; Men; Women; San Diego; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Multiple Endocrine Neoplasia Type 1; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pistachio-enriched diet (Experimental): Participants in this group will be individually counseled on a lower calorie diet, receive pistachios to be consumed daily for four months, and receive print materials on incorporating pistachios into their diet.
  Interventions: Behavioral: Pistachio-enriched diet
- General dietary guidance diet (Active Comparator): Participants in this group will receive general dietary guidance as part of a 4-month long group intervention.
  Interventions: Behavioral: General dietary guidance diet

INTERVENTIONS:
Behavioral: Pistachio-enriched diet — Composition of prescribed diets will be based on individual preferences, with the goal of consuming 1.5 oz of pistachios per day and increased energy expenditure. During the 4-month intervention, study subjects will participate in individualized counseling and group sessions, with in-person, telephone, email and text message contacts to provide support and behavioral guidance and strategies. Pistachios will be provided to participants. The overall content of the intervention consists of key elements of cognitive-behavioral therapy for obesity. The physical activity component emphasizes planned aerobic exercise, increased physical activity in the lifestyle, and strength training.
  Arms: Pistachio-enriched diet
Behavioral: General dietary guidance diet — During the 4-month group intervention, study subjects will participate group sessions, receive telephone, email and/or text message contacts to provide support and behavioral guidance and strategies. The overall content of the intervention consists of key elements of cognitive-behavioral therapy for obesity. The physical activity component emphasizes planned aerobic exercise, increased physical activity in the lifestyle, and strength training.
  Arms: General dietary guidance diet

SUMMARY:
The purpose of the Get Fit, Be Fit Study is to examine the effect of incorporating pistachios in an intensive 4-month cognitive-behavioral weight loss intervention in overweight and obese men and women, to examine effects on metabolic factors, and to monitor and examine changes in dietary intake and food choices during the intervention, in a randomized controlled study.

DETAILED DESCRIPTION:
This study investigates whether pistachios help to promote weight loss and improve metabolic and cardiovascular disease risk factors in 100 overweight or obese men and women who are participating in a 4-month behavioral weight loss intervention. Participants will be assigned to a cognitive-behavioral weight loss intervention and will be provided either general dietary advice as a component of the behavioral curriculum or prescribed an individualized pistachio-enriched reduced-energy diet plan. The pistachio-enriched diet will prescribe 42 g/day of pistachios, or approximately 13-20% (averaging 18%) of energy intake across a range of 1200-1800 kcal/day. Dietary intake will be assessed at three time points (baseline, one month, and four months) to examine changes in dietary intake and food choices that may be indicative of compensatory intake in response to regular nut consumption. Results from this study will contribute to understanding the role of pistachios in weight control, including further knowledge of the metabolic factors linked to chronic disease, and will expand knowledge of how pistachios in the diet may contribute to the prevention and management of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women who reside in the San Diego area
* Age 21 and older
* BMI ≥ 27.0 kg/m2 and ≤40 kg/m2
* No known allergy to tree nuts
* Non-diabetic
* Non-smoker
* Willing and able to participate in clinic visits, group sessions, and telephone and Internet communications at specified intervals
* Able to provide data through questionnaires and by telephone
* Willing to maintain contact with the investigators for 6 months
* Willing to allow blood collections
* Capable of performing a simple test for assessing cardiopulmonary fitness
* Willing and able to be physically active

Exclusion Criteria:

* Inability to participate in physical activity because of severe disability
* Inability to restrict consumption of nuts for four months
* History or presence of a co-morbid disease for which diet modification and increased physical activity may be contraindicated
* Self-reported pregnancy or breastfeeding or planning a pregnancy within the next year
* Currently actively involved in another diet intervention study or organized weight loss program
* Having a history or presence of a significant psychiatric disorder or any other condition that, in the investigator's judgment, would interfere with participation in the trial.
* Prior to enrollment
* Subjects will be screened for diabetes and considered ineligible with a fasting blood glucose ≥125 mg/dL.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 4 months
  Weight loss after a 4-month cognitive-behavioral intervention among the pistachio enriched diet arm as compared to general dietary guidance study arm.

SECONDARY OUTCOMES:
Metabolic and cardiovascular disease risk | 4 months
  The differential response in metabolic and cardiovascular disease risk factors, including lipids, glucose, insulin and insulin resistance among the pistachio enriched diet arm as compared to general dietary guidance study arm after four months.

OTHER OUTCOMES:
Dietary intake and food choices | 4 months
  The differential response in dietary intake and food choices in association with prescribing the pistachio-enriched diet as compared to general dietary guidance at 2-months and 4-months.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Rock, PhD, RD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No